CLINICAL TRIAL: NCT02456779
Title: Assessment of Equivalence of a Non-invasive In-vitro Diagnostic Test (Peptest) in Comparison to Other Routine Clinical Diagnostic Methods for GERD by Testing a Large Number of Clinical Samples
Brief Title: Validation of a Non-invasive In-vitro Diagnostic Test (Peptest) Against Other Diagnostic Methods for GERD
Acronym: PEPTESTCN
Status: Completed | Type: Observational
Sponsor: MAAB (Shanghai) Medical Device Limited (Industry)
Collaborators: RD Biomed Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: PEPTESTCN
Record Dates: First submitted 2015-05-21; First posted 2015-05-29 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Gastro-esophageal Reflux Disease
Keywords: pepsin; peptest; GERD; NERD; diagnostic
MeSH Terms: conditions — Gastroesophageal Reflux; Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples will be obtained from each subject. Specimens will be disposed of after testing for presence of pepsin using Peptest.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Erosive Esophagitis: Patients diagnosed with GERD with erosive esophagitis present on routine endoscopy during the previous 6 months.
  RDQ greater or equal to 12
  Saliva samples to be obtained intervention: in vitro diagnostic test Peptest intervention: questionnaire
  Interventions: Other: in vitro diagnostic test (Peptest); Other: Questionnaire
- non erosive reflux disease: Patients diagnosed with GERD with erosive esophagitis not present on routine endoscopy during the last 6 months.
  RDQ greater or equal to 12
  Saliva samples to be obtained intervention: in vitro diagnostic test Peptest intervention: questionnaire
  Interventions: Other: in vitro diagnostic test (Peptest); Other: Questionnaire
- healthy controls: No GERD symptoms RDQ = 0 RSI = 0-9
  Saliva samples to be obtained intervention: in vitro diagnostic test Peptest intervention: questionnaire intervention: questionnaire
  Interventions: Other: in vitro diagnostic test (Peptest); Other: Questionnaire

INTERVENTIONS:
Other: in vitro diagnostic test (Peptest) — saliva samples obtained and tested in laboratory conditions for the presence of pepsin using Peptest
  Other Names: Peptest
Other: Questionnaire — all recruited subjects to complete the RDQ as a determinant of inclusion criteria
  Other Names: Reflux Disease Questionnaire (RDQ)
Other: Questionnaire — control subjects to complete RSI as a determinant of inclusion criteria
  Other Names: Reflux Symptom Index
  Groups: healthy controls

SUMMARY:
The primary objective of this clinical study is to determine whether Peptest (Human Pepsin lateral flow in vitro diagnostic medical device) is equivalent to other GERD diagnostic methods commonly applied in clinical practice by testing a large number of clinical samples.

This will be performed by evaluating Peptest results in GERD patients (Erosive esophagitis or NERD), defined using standard clinical procedures, and compared to healthy controls.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) mainly manifests as three types, erosive esophagitis (EE), non-erosive reflux disease (NERD) and Barrett's esophagus. EE is characterized by damaged distal esophageal mucosa which is visible by endoscope, and also referred to as "endoscopically positive gastroesophageal reflux disease". NERD is defined as discomfort related to reflux without any obvious mucosal damage by endoscope, and is also known as "endoscopically negative gastroesophageal reflux disease".

At present the diagnosis of GERD uses syndrome-based diagnosis, proton pump inhibitor (PPI) test, 24-hour esophageal pH monitoring, endoscopy, etc. However, some of the above methods lack specificity and some may bring great suffering to patients due to being invasive (e.g., 24-hour esophagus pH monitoring). The disadvantage of endoscopy lies in its low detection rate, only 2.95% to 4.1% as NERD is the most frequent diagnosis. Therefore, diagnosis based on GERD syndromes still remains one of the most common diagnostic methods. In recent years, questionnaire surveys about GERD have been carried out at abroad, aiming at finding a simple and feasible diagnostic method. As one of the worlds's most recognized and commonly used diagnostic scale for the diagnosis of GERD, reflux disease questionnaire (RDQ) is a survey of medical history mainly based on symptom score. Studies at both home and abroad have confirmed its validity and reliability in the diagnosis of GERD. The reflux symptom index (RSI) is a validated questionnaire used to confirm the presence (or absence) of extra-esophageal reflux that are atypical symptoms of reflux that control subjects may overlook.

Peptest (Human Pepsin lateral flow in vitro diagnostic medical device) can be used in clinic for fast and convenient pepsin detection in patients' saliva. Pepsin, detected from saliva samples, can be regarded as a marker of a reflux event for the diagnosis of gastroesophageal reflux disease.

The primary objective of this study is to determine whether Peptest (Human Pepsin lateral flow in vitro diagnostic medical device) produced by RD Biomed Limited is equivalent to other GERD diagnostic methods commonly applied in clinical practice by testing a large number of clinical samples.

GERD patients and controls will provide saliva samples and these will be tested for the presence of pepsin using Peptest. Peptest results (positive or negative) will be evaluated in GERD patients (Erosive esophagitis or NERD) defined using standard clinical diagnostic tools and compared to controls (confirmed to not have reflux using two validated questionnaires).

ELIGIBILITY:
Inclusion Criteria:

Case group:

* Patients diagnosed as gastroesophageal reflux disease within 6 months had endoscopy within 6 months and presented with reflux symptoms in the past 4 weeks.
* Patients with RDQ questionnaire score of no less than 12 points.
* Patients who met the requirements and signed the informed consent.
* Collection and processing of samples should comply with the requirements of laboratory operation rules and product specifications.

Healthy group:

* Healthy subjects without any symptoms of gastroesophageal reflux, extra-esophageal reflux and laryngopharyngeal reflux.
* Healthy subjects with RDQ questionnaire score of 0.
* Healthy subjects with RSI questionnaire score of no more than 9 points and heartburn symptom score of 0.
* Healthy subjects who met the requirements and signed the informed consent.
* Collection and processing of samples should comply with the requirements of laboratory operation rules and product specifications.

Exclusion Criteria:

* Patients with functional heartburn.
* Patients who took gastric motor drugs within 7 days after entering the study.
* Patients with esophageal spasm and achalasia, eosinophilic esophagitis, dysphagia, esophageal or gastric cancer, and patients who received esophagus and stomach surgery
* Patients with serious hypohepatia or renal insufficiency
* Pregnant women
* Patients whose saliva samples were not appropriate for detection
* Samples not meeting the collection and processing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: GERD patients Erosive Esophagitis (EE) Non-erosive reflux disease (NERD) Heathly controls with GERD symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Peptest result (+ or -) | baseline
  Proportion of GERD patients Peptest positive compared to controls that are Peptest postitive

SECONDARY OUTCOMES:
Peptest result (+ or -) | baseline
  Proportion of EE, NERD patients and control Peptest positive
Peptest result (+ or -) | baseline
  Proportion of GERD patients Peptest positive within 15 minutes of symptoms
Peptest result (+ or -) | baseline
  Proportion of Peptest positive in comparison to reference diagnostic test
Safety (adverse events) | baseline
  adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yuan Fang, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (9):
- China (9):
  - Beijing Jishuitan Hospital, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Huadong Hospital afflicted to Fudan University, Shanghai
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Ruijin Hospital, School of Medicine, Shanghai Jiaotong University,, Shanghai
  - Shanghai East Hospital Affiliated to Tongji University, Shanghai
  - The Shanghai Tenth People's Hospital of Tongji University, Shanghai
  - Tongji Hospital, Tongji University School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai